CLINICAL TRIAL: NCT02165579
Title: Osteomyelitis: Procalcitonin to Diagnose and Monitor Osteomyelitis
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Biomarkers for Osteomyelitis
Record Dates: First submitted 2014-05-12; First posted 2014-06-17 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Diabetes; Foot Ulcer; Osteomyelitis
Keywords: procalcitonin; biomarkers; Osteomyelitis; diabetes; foot ulcer(s); Infectious Disease Society of America stage 3 infection
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Osteomyelitis | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Age > 21, diabetes, osteomyelitis: 1 Cohort, standard care, observational patients are: Diagnosis of diabetes mellitus Age ≥ 21 years Infectious Disease Society of America stage 3 infection
  Interventions: Other: 1 cohort, standard care, observational

INTERVENTIONS:
Other: 1 cohort, standard care, observational — This is one cohort standard care observational study. 40 diabetic patients admitted to Parkland hospital with a foot infection. We will enroll a representative cross section of subjects with diabetic foot infection. Patient will be consented and will receive therapy based on standard protocols. Currently patients with suspected osteomyelitis have bone biopsies to identify bacterial pathogens and verify MRI diagnosis. Repeat bone biopsies are performed at the end of therapy to verify that osteomyelitis has been successfully treated. Serum to measure procalcitonin will be obtained at baseline, week 3 and week 6. Tissue samples will be obtained at Baseline, Week 3 and Week 6 for tissue culture.

SUMMARY:
The investigator plans a cohort study of 80 subjects admitted to hospital with a diabetic foot infection in order to compare serial bone biopsies (the current "gold standard") and procalcitonin to diagnose and monitor the effectiveness of therapy for osteomyelitis. The investigator will collect specimens as part of an existing trial to evaluate negative pressure wound therapy in diabetic infected wounds. A high proportion of these patients have osteomyelitis and will receive standard therapy including repeat bone biopsy and parenteral antibiotics. The investigator expects repeated measurement of procalcitonin will be highly correlated with repeated bone biopsy after antibiotic treatment has been completed to determine if therapy has been successful or if additional antibiotic therapy is needed.

DETAILED DESCRIPTION:
There is a world-wide epidemic of diabetes. As part of the epidemic lower extremity amputations are dramatically increasing. Soft tissue and bone infections are one of the most common reasons for amputation. It is often difficult to determine if diabetic foot ulcers have an underlying bone infection. Inaccurate diagnosis of osteomyelitis leads to unnecessary antibiotic treatment, surgery, and amputation. In addition, we do not have good diagnostic tools to determine when osteomyelitis has been treated successfully.

The role of biomarkers specific to bone turnover (resorption and formation) in relation to bone infections is poorly understood. We know that remodeling is an essential function in bone physiology with increased osteoclast production leading to resorption of old bone coupled with increased osteoblast production associated with new bone formation. The balance between these two functions is known to be disrupted in disease states including osteoporosis, but has not been examined specifically in infected bone. Procalcitonin has been suggeasted as a tool to both diagnose and monitor the effectiveness of therapy for various infections, but there is very little work in diabetic foot osteomyelitis.

Aim 1. To evaluate the role of procalcitonin as a screening tool to diagnose diabetic foot osteomyelitis using bone culture and histopathology as the "gold standard" to establish the diagnosis.

Aim 2. To determine the role of procalcitonin as a management tool to determine osteomyelitis treatment success versus treatment failure (indicated by bone biopsy) after completing a standard course of antibiotics for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Age ≥ 21 years
* Infectious Disease Society of America stage 3 infection

Exclusion Criteria:

* History of previous bone infection in the study foot
* Unable to provide informed consent
* HIV, Hepatitis, osteomyelitis at other sites

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age > 21, diabetes, Infectious Disease Society of America stage 3 infection (osteomyelitis)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
(1.) wound healing, | 6 months
  Clinical examination. Per current standards, wound healing will be defined as complete granulation over the wound bed (primary intention) or wounds closed by surgical intervention. 80 subjects will be followed during the course of the study and the wound healing dates recorded for those subjects who heal.

SECONDARY OUTCOMES:
(2.) limb salvage | 6 months
  Clinical examination. This outcome will be measured by the number of subjects not requiring amputation during the time frame of the study.
(3.) hospitalizations for recurrent diabetic foot infection | 6 months
  The medical record will be reviewed on each subject and dates of hospitalizations for diabetic foot infection will be recorded.
(4.) surgical procedures | 6 months
  The medical record will be reviewed for each subject, and the dates and surgical procedures will be recorded.
(5.) recurrent ulcers. | 6 months
  The medical record will be reviewed for each subject and any recurrence of diabetic foot ulcers during the time frame of the study will be recorded. Data will include the date(s) of recurrence, location and size of the ulcer(s), and the presence or absence of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States